CLINICAL TRIAL: NCT06243354
Title: An Open-label, Multi-center, Multi-cohort, Phase 1/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HYP-2090PTSA in Patients With Advanced Solidt Tumors Harboring KRAS Mutation
Brief Title: Phase 1/2 Study of HYP-2090PTSA in Patients With Advanced Solid Tumors Harboring KRAS Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY0002-101
Record Dates: First submitted 2024-01-25; First posted 2024-02-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Safety; Tolerability; Efficacy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test product-HYP-2090PTSA (Experimental)
  Interventions: Drug: Test product: HYP-2090PTSA

INTERVENTIONS:
Drug: Test product: HYP-2090PTSA — Dosage form: Capsule. Strength: 2.5 mg, 5 mg and 10mg. Method of administration: Take orally on an empty stomach. Do not chew. Swallow the product with warm water.
  Dose Escalation Phase PK Lead-in Period (C0D1 only): Take once (QD dosing regimen only). Starting from C1D1, and in the Dose Expansion part, subjects will take the protocol-specified dose of HYP-2090PTSA orally in the morning on an empty stomach and one hour before the evening meal (evening dosing applies to BID regimen only), administered once to twice daily or two to three times per week. The administration dosages are: QD (once daily); BID (twice daily); TIW (on Days 1, 3, and 5 of each week); BIW (on Days 1 and 4 of each week).
  Avoid drinking water as much as possible within 1 hour before and after dosing (except for the water taken with the medication).
  Do not re-administer the dose if vomiting occurs after drug intake.

SUMMARY:
This is a multicenter, open-label phase 1/2 study consisting of two parts: dose escalation phase and dose expansion phase. The objective of the dose escalation phase is to evaluate the safety, tolerability and pharmacokinetics of HYP-2090PTSA in patients with advanced solid tumors harboring KRAS mutation and to determine the RP2D. In the dose expansion phase, preliminary efficacy and safety at the RP2D will be further explored in patients with specific cancer harboring KRAS p.G12C mutation.

ELIGIBILITY:
Inclusion Criteria:

* A written informed consent should be signed by a subject or his/her legal representative before any study-related procedures are performed;
* 18 Years and older;
* Subjects with histologically or cytologically confirmed locally advanced or metastatic advanced solid tumors;
* Subjects must have at least one measurable lesion as defined by RECIST v1.1;
* Eastern Cooperative Oncology Group(ECOG) performance status 0-1;
* Expected survival ≥ 3 months;
* Patients are willing to use a highly effective method of birth control during the study, and for at least 180 days after the last dose of study medication.

Exclusion Criteria:

* Patients who have received major surgical or interventional treatment within 4 weeks prior to the first dose, with the exception of tumor biopsy, puncture, etc. Patients who have received anti-tumor therapy (radiotherapy, immunologic therapy or biological therapy) within 4 weeks, prior to the first dose, or received small molecular targeted therapy, chemotherapy within 2 weeks, or received palliative radiotherapy for bone metastases within 2 weeks, or received nitrosoureas or mitomycin C within 6 weeks;
* Patients who have received live vaccines within 4 weeks prior to the first dose;
* Patients who have previously participated in clinical trials of other drugs within 4 weeks before the first dose;
* Patients with a history of central nervous system disease within 12 months prior to enrollment, such as seizures, cerebral vascular embolism/hemorrhage, paralysis, aphasia, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, psychiatric disease, or any autoimmune disease with involvement of the central nervous system;
* Presence of severe pulmonary diseases such as pulmonary embolism, interstitial lung disease at screening;
* Patients who have previously received allogeneic tissue/solid organ transplantation;
* Patients with active infection;
* Patients who are positive for human immunodeficiency virus (HIV) (HIV1/2 antibody), positive treponema pallidum antibody (positive treponema pallidum antibody is required to undergo a confirmatory test, and those with negative confirmatory test can be enrolled), active chronic hepatitis B (HBsAg positive and HBV DNA > 500 IU/mL) or active hepatitis C (HCV antibody positive and HCV-RNA > lower limit of detection by the research center);
* Female subjects who are lactating or have a positive blood/urine pregnancy result during the screening period;
* Any other condition of the subject (e.g., mental, geographical, or medical condition) that does not allow him or her to comply with the study and follow-up procedures, or other conditions that, in the judgment of the investigator, the subject is not suitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recommended phase-2 dose (RP2D) | Approximately 2 years
  RP2D should be selected based on a comprehensive assessment of maximum Tolerated dose (MTD), toxicity, pharmacokinetic (PK) profile, and efficacy data
Number of participants with dose limiting toxicities | 24 days
  Dose-limiting toxicity (DLT) is defined as an adverse event (AE) or clinically Significant abnormal laboratory value occurring in DLT assessment period

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Approximately 2 years
  All patients participating in this study will be assessed for incidence and severity of AEs and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imagings and ophthalmological assessments
Objective response rate (ORR) | Approximately 2 years
  ORR is defined as the proportion of participants with confirmed complete response or partial response
Progression-free survival (PFS) | Approximately 2 years
  Period of time from the start of treatment to tumor progression or death from any cause (whichever occurs first) based on RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Hunan Provincial Cancer Hospital, Changsha, Hunan
  - The first Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Provincial Cancer Hospital, Jinan, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided